CLINICAL TRIAL: NCT03267277
Title: An Open-label Study of Sodium Thiosulfate for Treatment of Calcinosis Associated With Juvenile and Adult Dermatomyositis
Brief Title: Sodium Thiosulfate for Treatment of Calcinosis Associated With Juvenile and Adult Dermatomyositis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170161; 17-E-0161 (Other: NIHCC)
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Results first posted 2024-02-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2022-10

CONDITIONS: Dermatomyositis; Idiopathic Inflammatory Myopathies
Keywords: Calcinosis; Dermatomyositis; Juvenile Dermatomyositis; Idiopathic Inflammatory Myopathies; Sodium Thiosulfate
MeSH Terms: conditions — Dermatomyositis; Myositis; Calcinosis | interventions — sodium thiosulfate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants received intravenous sodium thiosulfate 16 g/m^2 three times weekly for 10 weeks
  Interventions: Drug: Sodium Thiosulfate

INTERVENTIONS:
Drug: Sodium Thiosulfate — Sodium thiosulfate is a calcium chelator

SUMMARY:
Background:

Dermatomyositis (DM) and juvenile dermatomyositis (JDM) cause inflammation in the muscles. People with DM and JDM can develop calcium deposits in places they should not, known as calcinosis. Calcinosis can be painful and cause disabilities and other problems. Researchers want to learn more about calcinosis to find treatments for it.

Objective:

To test if sodium thiosulfate (STS) can treat people with DM with calcinosis.

Eligibility:

People ages 7 and older who have moderate or severe calcinosis. They must have stable DM and calcium deposits in the torso or at least 2 limbs.

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Muscle strength and function tests
* Blood and urine tests

Participants will have several visits:

* 7-day pre-treatment visit about 10 weeks before starting STS
* Treatment visits over 10 weeks. They will get STS 3 times a week through IV infusion. They may be hospitalized the whole time. If they tolerate the drug, they may be discharged at certain times. During these times, they will return for the infusions.
* 3- to 5-day post-treatment visits 24 weeks and 62 weeks after starting STS.

Visits may include repeats of screening tests and:

* Questionnaires
* Scans: They lie in a machine that takes pictures of the body. They may be injected with a radioactive agent.
* Durometry: A small instrument applies pressure on the skin or exposed calcinosis.
* Measurements of blood flow in the arms and fingernail blood vessels
* Photographs of the skin
* Kidney ultrasound
* Tests of kidney function
* Calcinosis aspiration: A needle placed into areas of calcinosis removes liquid.

DETAILED DESCRIPTION:
Calcinosis, a serious complication of dermatomyositis, involves deposition of calcium (carbonate apatite) in soft tissue, and can result in negative impacts on quality of life and physical function. To date, there are no known effective therapies that are approved for the treatment of dermatomyositis-associated calcinosis, and there is no consensus within the medical community on the optimum treatment strategy for this often-debilitating condition.

A few reports in the literature describe treatment successes with a variety of therapeutics; however, these data are from anecdotal reports or case series and thus provide limited scientific evidence of effectiveness. Recently published reports as well as personal observations within our group have suggested that intravenous sodium thiosulfate treatment may benefit calcinosis patients. In order to gather more robust data on the utility of this medication in the treatment of calcinosis associated with adult and juvenile dermatomyositis, we propose to evaluate its effects in the context of a prospective clinical trial.

We plan to enroll participants at a single center into a single-arm, open-label study, with the overall objective of evaluating the efficacy and safety of intravenous sodium thiosulfate use in patients with moderate to severe extensive calcinosis associated with juvenile and adult dermatomyositis.

The study will enroll a maximum of 18 participants over 4 years into the full study, but up to 250 patients may screen for study entry. Eligible patients will be age 7 or older, and will have extensive calcinosis (defined as calcinosis involving the torso or 2 extremities) and moderate to severe calcinosis (indicated by a calcinosis activity visual analogue scale score of greater than or equal to 3.5 cm out of 10 cm).

Two separate evaluations performed at the NIH prior to initiation of therapy will be used as baseline data to compare in a pairwise manner to the change in assessments following treatment with sodium thiosulfate, with all other medications remaining stable. Study treatment will be 16 g/m2 sodium thiosulfate administered 3 times weekly over a period of 10 weeks at the NIH. Subjects who complete 10 weeks of treatment or reach the primary end point by week 6 will be considered completers. Following the treatment period, all participants will return to the NIH for evaluations at weeks 24 and 62.

The primary outcome will be change in calcinosis activity visual analogue scale score from week 0 to week 10 on therapy, compared to the baseline change in calcinosis activity visual analogue scale score from week -10 to week 0 pre-treatment. Secondary measures will evaluate safety and changes in components of the Calcinosis Assessment Tool, clinical assessments of calcinosis, Mawdsley Calcinosis Questionnaire, quality of life, functional disability, muscle testing (manual and quantitative), laboratory parameters (muscle enzymes, inflammatory markers, and endothelial activation markers), gene expression, calcification pathogenesis, time to improvement, and imaging. Myositis disease activity and damage will also be assessed by validated measures.

A number of research studies will be incorporated into this clinical trial in an attempt to understand the immunologic markers associated with calcification in dermatomyositis as well as the immunologic effects of sodium thiosulfate treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. At least 7 years of age
  2. Meets Bohan and Peter criteria, as modified by the International Myositis Assessment and Clinical Studies Group (IMACS), for probable or definite DM or JDM
  3. Has extensive calcinosis, defined as calcinosis involving at least 2 extremities or the torso
  4. Has moderate to severe calcinosis, defined as having a calcinosis activity visual analogue scale score of greater than or equal to 3.5 cm out of 10 cm
  5. Is willing and able to comply with the requirements of the protocol and to undergo all testing
  6. Can have IV access established to receive study infusions
  7. Myositis disease activity is stable*
  8. Medications for myositis are stable for at least 6 weeks prior to study entry**
  9. Men and women of reproductive potential must agree to use a reliable form of birth control during the 62-week duration of the study
  10. Subjects or their legal guardian must sign a written informed consent

      * Stable myositis disease activity will be defined by physician global and patient/parent global VAS that are <4 cm, as well as creatine kinase (CK), lactate dehydrogenase (LDH), aldolase, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) that are less than or equal to 2X upper limit of normal (ULN).

        * If a patient has a medication for myositis changed in this window for reasons besides their myositis activity and has returned to their baseline medication use prior to enrollment they will still be eligible.

EXCLUSION CRITERIA:

1. Is pregnant or breastfeeding
2. Has known allergies to sodium thiosulfate, any of its components, or dextrose
3. Has severe myositis disease activity as defined by patient/parent or physician global activity visual analogue scale score >4 cm out of 10 cm
4. Has had an escalation of immunosuppressive therapy in the 2 months prior to enrollment for the purpose of treating active myositis disease activity, including the addition of a new agent to treat the patients underlying disease or an increase in dose of an existing medication used to treat the patient's disease (other than an adjustment for weight or body surface area in children)
5. Has a malignancy or had a malignancy within 5 years of diagnosis of their DM (except for benign skin lesions or basal cell carcinoma)
6. Known or suspected history of alcohol or drug abuse in the 6 months prior to study enrollment
7. Has systemic lupus erythematosus, scleroderma, or a condition other than DM that is associated with calcinosis as a complication
8. Has had a change in medications used specifically for calcinosis in the 2 months prior to enrollment, including but not limited to alendronate, etidronate, pamidronate, probenecid, colchicine, diltiazem, thalidomide, and aluminum hydroxide
9. Has used probenecid, diltiazem, aluminum hydroxide, or hydrochlorothiazide in the 2 months prior to enrollment
10. Has currently or has a history of any of the following: heart failure, renal impairment (GFR less than 30 representing severe renal disease), liver disease (Child-Pugh class C), arrhythmias (that are symptomatic or are concerning for progression to symptomatic arrhythmias), or recurrent kidney stones (more than one episode of symptomatic kidney stones separated by at least 1 month), or QT prolongation, or hypocalcemia, or metabolic acidosis, or hypotension
11. Has severe osteoporosis or has had a bone fracture within a year prior to enrollment. For adults, severe osteoporosis as defined by the World Health Organization (WHO) as bone mineral density (BMD) 2.5 standard deviations below that of a young, normal adult (T-score at or below -2.5 and one or more fractures). For individuals, less than age 18, severe osteoporosis as defined by the First Pediatric Consensus Development Conference as a Z-score below -2 and one or more fractures.
12. Has a psychiatric illness or medical non-compliance that the study team feels will make the patient unlikely to complete the study
13. Has dysphagia where non-oral feeding alternatives are needed.
14. Requires supplemental oxygen therapy
15. Has >3 episodes of cellulitis requiring IV antibiotics related to calcinosis within a year prior to enrollment or cellulitis within 1 month of enrollment
16. Previously received or currently receiving sodium thiosulfate by any route
17. Is on an oral prednisone dose of more than 1mg/kg/day or other oral corticosteroid equivalent.
18. Is taking any concomitant medications that are thought to alter sodium thiosulfate s effects or pharmacokinetics. Once patients have met all other inclusion criteria and no other exclusion criteria this criteria will be checked. A PharmD will evaluate the patient's current medication list for medications with the potential for interaction with sodium thiosulfate. Methodology is as follows: He or she will perform a search in two individual validated medication interaction software programs. He or she will also perform a literature search via PubMed for case reports of interactions with sodium thiosulfate. As an additional safeguard, the PharmD will evaluate the medication list utilizing principles of pharmacology and pharmacokinetics to attempt to identify any potential interactions not yet documented in the literature.
19. Has any health conditions that, in the opinion of the investigator, significantly increase the risk of taking sodium thiosulfate or participating in any of the study procedures
20. Weighs less than 26 kilograms.**
21. Has a regimen of pulse steroids or intravenous immunoglobulin (IVIG) that is at an interval besides every 1, 2, or 5 weeks.
22. Has a chronic infection that makes assessment of muscle disease difficult including, but not limited to, hepatitis, HIV, HTLV 1, and HTLV 2.
23. Has had a severe complication of diabetes in the past year prior to enrollment.
24. Anemia with a hemoglobin (HgB) less than 10 at time of screening or deemed to be too low to safely complete study by hematology consult team.
25. We will attempt to enroll patients at a weight greater than 28 kg as these patients will be able to obtain all lab work for the study. Patients weighing 26 to 28 kg will only be able to obtain some of the research blood work. Patients less than 26 kg of body weight will be unable to obtain all safety labs, so will not be able to enroll.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam I Schiffenbauer, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-E-0161.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 participants were consented but one participant was a screen failure so was not enrolled to the treatment phase of the study.
Period: Overall Study
Arm/Group | Treatment
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 7
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Calcinosis Activity Visual Analogue Scale Score
Description: Calcinosis activity is defined by the metabolic activity and the inflammation associated with calcinosis. In evaluating calcinosis activity, the study physicians take into account the change in extent of calcinosis and the location of calcinosis lesions, the consistency and texture of calcinosis lesions, the presence of erythema surrounding calcinosis lesion, and any pain associated with the calcinosis lesions. A 10 cm visual analogue scale (VAS) was scored by a physician with a vertical line on the scale marking calcinosis activity where 0 cm indicates no evidence of calcinosis, and 10 cm mark indicates severe calcinosis activity. The change in calcinosis activity VAS score from week 0 to week 10 on therapy was compared to the change in calcinosis activity VAS score from week -10 to week 0 on baseline therapy. The baseline score was calculated by taking the week 0 score minus the week -10 score. The on therapy score was calculated by taking the week 10 score minus the week 0 score.
Time Frame: Week 10 minus week 0 (on therapy) and week 0 minus week -10 (baseline)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 13
Units on a scale | -3.45 (0.89)

2. Secondary Outcome: Change in Quality of Life Measured by the Child Health Questionnaire-Parent Form 50 (CHQ-PF50): Physical Function Domain
Description: The Child Health Questionnaire-Parent Form 50 (CHQ-PF50) is a 50-item survey with 14 domains that parents complete to assess their child's physical and mental well-being. The change in quality of life was measured by the physical functioning domain score on the CHQ-PF50. The CHQ-PF50 physical functioning domain scale was transformed to 0 to 100 score with higher score indicating better health or more positive functioning. The change in quality of life using the CHQ-PF50 score was measured as the mean difference in scores between time points.
Time Frame: Week -10 to 0 (pre-treatment); Week 0 to 10 (on treatment)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 13
Units on a scale
  Pre-treatment | -1.00 (6.15)
  On treatment | -8.00 (11.60)

3. Secondary Outcome: Change in Quality of Life Measured by the 36-Item Short Form Health Survey (SF-36) Score: General Health Domain
Description: 36-Item Short Form Health Survey (SF-36) is a 36-item patient-reported survey of patient health status that consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The Change in quality of life measured was assessed using the general health domain of SF-36. The higher the score the less disability. The change in quality of life using the SF-36 general health domain was measured as the mean difference in scores between time points.
Time Frame: Week -10 to 0 (pre-treatment); Week 0 to 10 (on treatment); Week 24 to 62 (post-treatment)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 13
Units on a scale
  Pre-treatment | 2.50 (7.17)
  On treatment | -1.00 (6.15)
  Post treatment | -8.00 (11.60)

4. Secondary Outcome: Improvement of Calcinosis Lesions Measured by the Change in Mawdsley Calcinosis Questionnaire (MCQ) Score
Description: The Mawdsley Calcinosis Questionnaire (MCQ) is a 17-item questionnaire scale that measures the severity and impact of calcinosis. Each item is scored on 11-point scale of 0 to 10. Total score is the the average of the cumulative measure ranging from 0-10. Higher score indicates worse severity and impact of calcinosis. Improvement of calcinosis lesions was measured by the MCQ. The change in score was measured as the mean difference between time points.
Time Frame: Week -10 to 0 (pre-treatment); Week 0 to 10 (on treatment); Week 24 to 62 (post-treatment)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 13
Units on a scale
  Pre-treatment | 0.33 (1.54)
  On treatment | -0.74 (2.18)
  Post treatment | -0.17 (0.86)

5. Secondary Outcome: Change in Quality of Life Measured by Skindex-29 Score
Description: The Skindex-29 scale is 29-item questionnaire that measures the quality of life. Each item is scored 0 (Never) to 4 (All the time). All responses are transformed to a linear scale of 100, varying from 0 (no effect) to 100 (effect experienced all the time) and overall score is the mean of the responses. Higher score indicates more severe impact on quality of life. The change in quality of life was measured as the mean difference in Skindex-29 scores between time points.
Time Frame: Week -10 to 0 (pre-treatment); Week 0 to 10 (on treatment); Week 24 to 62 (post-treatment)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 13
Units on a scale
  Pre-treatment | 1.77 (6.30)
  On treatment | -8.15 (10.63)
  Post treatment | -0.38 (6.53)

6. Secondary Outcome: Change in Muscle Strength Over Time Measured by Manual Muscle Test-8 (MMT-8) Score
Description: Manual Muscle Test-8 (MMT-8) is a measure of muscle strength. The MMT-8 uses a 10-point scale to score each muscle group, with 0 indicating extreme weakness and 10 indicating normal strength. The scores for each muscle group are then added together to get a total score ranging from 0 to 80, with higher scores indicating greater muscle strength. Change in muscle strength over time was measured as the mean difference in MMT-8 scores between time points.
Time Frame: Week -10 to 0 (pre-treatment); Week 0 to 10 (on treatment); Week 24 to 62 (post-treatment)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 13
Units on a scale
  Pre-treatment | -0.08 (3.40)
  On treatment | 1.38 (2.79)
  Post treatment | -0.27 (3.29)

7. Secondary Outcome: Change in Muscle Strength Over Time Measured by Quantitative Muscle Assessment (QMA): Hip Abductor Muscle
Description: Quantitative muscle assessment (QMA) tests how much force participant can be exerted by the hip abductor muscle. It is measured as the kilograms of force produced. Higher score indicates more force. Change in hip abductor muscle strength over time was measured by the quantitative muscle assessment (QMA) as the mean difference in QMA scores between time points.
Time Frame: Week -10 to 0 (pre-treatment); Week 0 to 10 (on treatment); Week 24 to 62 (post-treatment)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Treatment
Number analyzed (Participants) | 13
Kilograms
  Pre-treatment | 0.16 (1.26)
  On treatment | 0.74 (1.75)
  Post treatment | 1.35 (1.77)

8. Secondary Outcome: Change in Myositis Activity Measured by Physician Global Activity (PGA)
Description: The Physician Global Activity (PGA) is an index that uses a 10-cm Visual Analog Scale (VAS) to score a patient's disease activity. Higher score indicates more activity. Change in myositis activity was measured as the mean difference in disease activity scores between time points.
Time Frame: Week -10 to 0 (pre-treatment); Week 0 to 10 (on treatment); Week 24 to 62 (post-treatment)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 13
Units on a scale
  Pre-treatment | 0.36 (1.54)
  On treatment | -0.87 (1.27)
  Post treatment | -0.32 (0.47)

9. Secondary Outcome: Change in Myositis Damage Measured by Physician Global Damage (PGD)
Description: The Physician Global Damage (PGD) is an index that uses a 10-cm Visual Analog Scale (VAS) to score a patient's disease damage. Higher score indicates more global damage. Change in myositis damage was measured as the mean difference in disease damage scores between time points.
Time Frame: Week -10 to 0 (pre-treatment); Week 0 to 10 (on treatment); Week 24 to 62 (post-treatment)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 13
Units on a scale
  Pre-treatment | -0.02 (1.09)
  On treatment | -1.07 (1.09)
  Post treatment | -0.18 (0.53)

10. Secondary Outcome: Change in Total Percent Body Surface Area (BSA) Involved With Calcinosis
Description: Total percent of body surface area (BSA) involved with calcinosis was measured by physician assessment. Improvement of calcinosis lesions was measured as the mean difference in total percent of BSA scores between time points
Time Frame: Week -10 to 0 (pre-treatment); Week 0 to 10 (on treatment); Week 24 to 62 (post-treatment)
Population: The analysis only included those participants who completed 10 weeks of treatment
Measure: Mean (Standard Deviation); unit: percentage of Body Surface Area (BSA)
Arm/Group | Treatment
Number analyzed (Participants) | 13
percentage of Body Surface Area (BSA)
  Pre-treatment | 2.79 (4.06)
  On treatment | -10.18 (5.01)
  Post treatment | -0.45 (2.24)

ADVERSE EVENTS:
Time Frame: 62 weeks
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=14)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Catheter site infection (Infections and infestations) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1)
Calcium ionized decreased (Investigations) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=14)
Abnormal clotting factor (Blood and lymphatic system disorders) | 4 (8)
Anemia (Blood and lymphatic system disorders) | 13 (146)
Anisocytosis (Blood and lymphatic system disorders) | 2 (20)
Urine analysis abnormal (Blood and lymphatic system disorders) | 12 (336)
Sinus bradycardia (Cardiac disorders) | 4 (46)
Sinus tachycardia (Cardiac disorders) | 9 (280)
Dental caries (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (19)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hyperthermia (General disorders) | 2 (2)
Corona virus infection (Infections and infestations) | 3 (5)
Epstein-Barr virus infection (Infections and infestations) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (2)
Wound infection staphylococcal (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (5)
Activated partial thromboplastin time shortened (Investigations) | 6 (31)
Alanine aminotransferase (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (31)
Albumin urine present (Investigations) | 1 (4)
Aldolase increased (Investigations) | 4 (10)
Anion gap (Investigations) | 1 (1)
Anion gap decreased (Investigations) | 5 (20)
Anion gap increased (Investigations) | 5 (56)
Antinuclear antibody increased (Investigations) | 6 (6)
Antinuclear antibody positive (Investigations) | 3 (4)
Aspartate aminotransferase (Investigations) | 1 (1)
Aspartate aminotransferase decreased (Investigations) | 1 (13)
Aspartate aminotransferase increased (Investigations) | 5 (20)
Autoantibody positive (Investigations) | 2 (3)
Basophil count decreased (Investigations) | 3 (6)
Basophil count increased (Investigations) | 6 (13)
Basophil percentage increased (Investigations) | 7 (15)
Bilirubin urine present (Investigations) | 1 (1)
Blood albumin decreased (Investigations) | 10 (131)
Basophil percentage decreased (Investigations) | 3 (4)
Blood alkaline phosphatase decreased (Investigations) | 4 (60)
Blood bicarbonate decreased (Investigations) | 11 (103)
Blood bicarbonate increased (Investigations) | 11 (196)
Blood bilirubin decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Blood chloride decreased (Investigations) | 4 (29)
Blood chloride increased (Investigations) | 13 (73)
Blood cholesterol increased (Investigations) | 2 (3)
Blood creatine phosphokinase decreased (Investigations) | 1 (2)
Blood creatine phosphokinase increased (Investigations) | 6 (71)
Blood creatine phosphokinase MB increased (Investigations) | 4 (38)
Blood creatinine decreased (Investigations) | 9 (200)
Blood erythropoietin increased (Investigations) | 5 (8)
Blood folate increased (Investigations) | 2 (3)
Blood homocysteine increased (Investigations) | 1 (3)
Blood immunoglobulin A increased (Investigations) | 5 (67)
Blood immunoglobulin E increased (Investigations) | 6 (109)
Blood immunoglobulin D increased (Investigations) | 1 (1)
Blood immunoglobulin G increased (Investigations) | 10 (150)
Blood immunoglobulin M decreased (Investigations) | 3 (52)
Blood insulin increased (Investigations) | 5 (10)
Blood iron decreased (Investigations) | 6 (11)
Blood iron increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 13 (108)
Blood magnesium increased (Investigations) | 2 (5)
Blood parathyroid hormone (Investigations) | 1 (1)
Blood parathyroid hormone decreased (Investigations) | 1 (1)
Blood parathyroid hormone increased (Investigations) | 6 (10)
Blood phosphorus decreased (Investigations) | 7 (112)
Blood phosphorus increased (Investigations) | 6 (15)
Blood triglycerides increased (Investigations) | 3 (6)
Blood urea nitrogen decreased (Investigations) | 7 (97)
Blood urea nitrogen increased (Investigations) | 1 (31)
Blood uric acid increased (Investigations) | 4 (29)
Brain natriuretic peptide increased (Investigations) | 5 (15)
C-reactive protein-high sensitivity increased (Investigations) | 9 (67)
Calcium ionized decreased (Investigations) | 9 (53)
Calcium ionized increased (Investigations) | 4 (57)
Carbon dioxide decreased (Investigations) | 11 (142)
Carbon dioxide increased (Investigations) | 1 (1)
Citric acid urine decreased (Investigations) | 5 (13)
Citric acid urine increased (Investigations) | 1 (4)
Coagulation factor VIII level increased (Investigations) | 12 (32)
Creatinine urine decreased (Investigations) | 13 (270)
Creatinine urine increased (Investigations) | 9 (78)
Cystatin C increased (Investigations) | 8 (106)
Drug level above therapeutic (Investigations) | 1 (4)
Electrophoresis protein abnormal (Investigations) | 1 (1)
Eosinophil count decreased (Investigations) | 8 (21)
Eosinophil count increased (Investigations) | 1 (1)
Eosinophil percentage decreased (Investigations) | 6 (25)
Eosinophil percentage increased (Investigations) | 4 (18)
Fibrin D dimer increased (Investigations) | 1 (1)
Fibroblast growth factor 23 increased (Investigations) | 6 (8)
Flow cytometry (Investigations) | 14 (42)
Glucose urine present (Investigations) | 7 (133)
Glycosylated hemoglobin increased (Investigations) | 3 (5)
Immature granulocyte count increased (Investigations) | 10 (47)
Hemoglobin decreased (Investigations) | 1 (2)
Hemoglobin urine present (Investigations) | 6 (122)
Haptoglobin decreased (Investigations) | 1 (2)
Haptoglobin increased (Investigations) | 1 (1)
Hepatitis B core antibody positive (Investigations) | 3 (5)
Hepatitis B surface antigen positive (Investigations) | 3 (6)
Insulin C-peptide increased (Investigations) | 2 (2)
Low density lipoprotein abnormal (Investigations) | 1 (1)
Lymphocyte percentage decreased (Investigations) | 6 (10)
Lymphocyte percentage increased (Investigations) | 9 (35)
Mean cell hemoglobin decreased (Investigations) | 2 (12)
Mean cell hemoglobin increased (Investigations) | 1 (12)
Mean cell volume decreased (Investigations) | 1 (11)
Mean cell volume increased (Investigations) | 1 (15)
Mean platelet volume decreased (Investigations) | 6 (25)
Metamyelocyte percentage increased (Investigations) | 2 (5)
Monocyte percentage decreased (Investigations) | 6 (15)
Monocyte percentage increased (Investigations) | 3 (7)
Myelocyte percentage increased (Investigations) | 4 (5)
Neutrophil count decreased (Investigations) | 1 (1)
Neutrophil percentage decreased (Investigations) | 7 (20)
Neutrophil percentage increased (Investigations) | 6 (12)
Nitrite urine present (Investigations) | 2 (58)
PCO2 decreased (Investigations) | 11 (156)
PCO2 increased (Investigations) | 1 (1)
pH urine increased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 5 (24)
Platelet count increased (Investigations) | 2 (17)
Platelet morphology abnormal (Investigations) | 1 (1)
PO2 decreased (Investigations) | 3 (5)
PO2 increased (Investigations) | 11 (70)
Promyelocyte count increased (Investigations) | 1 (1)
Protein total decreased (Investigations) | 4 (33)
Protein total increased (Investigations) | 6 (75)
Protein urine present (Investigations) | 5 (57)
Prothrombin time shortened (Investigations) | 1 (2)
Red blood cell count decreased (Investigations) | 13 (140)
Red blood cell microcytes present (Investigations) | 1 (2)
Red blood cell morphology abnormal (Investigations) | 2 (8)
Red blood cell poikilocytes present (Investigations) | 1 (1)
Red blood cell sedimentation rate (Investigations) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 8 (22)
Red blood cells urine increased (Investigations) | 10 (84)
Red cell distribution width increased (Investigations) | 12 (134)
Reticulocyte count decreased (Investigations) | 1 (1)
Reticulocyte count increased (Investigations) | 6 (52)
Reticulocyte hemoglobin equivalent (Investigations) | 8 (23)
Reticulocyte percentage increased (Investigations) | 9 (47)
Serum ferritin decreased (Investigations) | 1 (1)
Serum ferritin increased (Investigations) | 7 (21)
Specific gravity urine increased (Investigations) | 2 (6)
T-lymphocyte count increased (Investigations) | 1 (3)
Transferrin increased (Investigations) | 1 (1)
Transferrin saturation increased (Investigations) | 1 (1)
Urinary casts present (Investigations) | 4 (14)
Urine albumin/creatinine ratio increased (Investigations) | 2 (3)
Urine calcium decreased (Investigations) | 5 (56)
Urine calcium increased (Investigations) | 3 (14)
Urine ketone body present (Investigations) | 10 (27)
Urine leukocyte esterase positive (Investigations) | 8 (128)
Urine magnesium decreased (Investigations) | 12 (38)
Urine magnesium increased (Investigations) | 7 (19)
Urine oxalate decreased (Investigations) | 6 (12)
Urine oxalate increased (Investigations) | 1 (1)
Urine phosphorus decreased (Investigations) | 10 (14)
Urine phosphorus increased (Investigations) | 6 (17)
Urine potassium decreased (Investigations) | 7 (68)
Urine potassium increased (Investigations) | 1 (1)
Urine protein/creatinine ratio increased (Investigations) | 12 (288)
Urine sodium decreased (Investigations) | 2 (2)
Urine sodium increased (Investigations) | 13 (36)
Urine uric acid decreased (Investigations) | 2 (4)
Urine uric acid increased (Investigations) | 4 (19)
Urobilinogen urine (Investigations) | 2 (4)
Venous oxygen saturation decreased (Investigations) | 14 (228)
Venous oxygen saturation increased (Investigations) | 14 (180)
Vitamin B12 increased (Investigations) | 2 (2)
Vitamin D decreased (Investigations) | 10 (29)
Vitamin D increased (Investigations) | 2 (4)
Von Willebrand's factor activity increased (Investigations) | 6 (15)
Von Willebrand's factor antigen increased (Investigations) | 4 (8)
White blood cell count decreased (Investigations) | 4 (18)
White blood cell count increased (Investigations) | 6 (22)
White blood cells urine increased (Investigations) | 12 (134)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (413)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 3 (8)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (146)
Hypoglycemia (Metabolism and nutrition disorders) | 9 (32)
Hypokalemia (Metabolism and nutrition disorders) | 13 (92)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (49)
Hyponatremia (Metabolism and nutrition disorders) | 13 (95)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Headache (Nervous system disorders) | 5 (21)
Anxiety (Psychiatric disorders) | 1 (1)
Urine amino acid level abnormal (Investigations) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 14 (422)
Hypotension (Vascular disorders) | 6 (95)
Absolute lymphocyte count decreased (Investigations) | 2 (17)
Absolute lymphocyte count increased (Investigations) | 5 (47)
Absolute monocyte count decreased (Investigations) | 4 (13)
Absolute monocyte count increased (Investigations) | 4 (19)
Absolute neutrophil count decreased (Investigations) | 4 (11)
Absolute neutrophil count increased (Investigations) | 7 (12)
Beta 2 microglobulin urine increased (Investigations) | 1 (1)
Bilirubin conjugated (Investigations) | 1 (1)
Human T-cell lymphotropic virus infection (Infections and infestations) | 3 (3)
Immature granulocyte percentage increased (Investigations) | 13 (71)
Ionized Magnesium decreased (Investigations) | 9 (87)
Ionized Magnesium increased (Investigations) | 9 (153)
Blood calcium decreased (Investigations) | 1 (13)
Blood creatinine increased (Investigations) | 1 (10)
Blood glucose increased (Investigations) | 1 (30)
Blood thyroid stimulating hormone decreased (Investigations) | 2 (6)
Blood thyroid stimulating hormone increased (Investigations) | 5 (18)
Catheter site infection (Infections and infestations) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 10 (47)
Creatinine renal clearance increased (Investigations) | 3 (9)
Cystatin C abnormal (Investigations) | 1 (20)
Diastolic hypertension (Vascular disorders) | 5 (30)
Diastolic hypotension (Vascular disorders) | 13 (448)
Erythroblast count increased (Investigations) | 7 (15)
Laboratory test (Investigations) | 1 (1)
Lipids abnormal (Investigations) | 1 (1)
Mean cell hemoglobin concentration decreased (Investigations) | 11 (86)
Migraine (Nervous system disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Procedural dizziness (Nervous system disorders) | 1 (1)
Prothrombin time prolonged (Investigations) | 2 (7)
Systolic hypertension (Vascular disorders) | 14 (515)
Thyroxine decreased (Investigations) | 1 (1)
Thyroxine free decreased (Investigations) | 2 (22)
Transferrin decreased (Investigations) | 2 (16)
Transferrin saturation decreased (Investigations) | 7 (13)
Urea renal clearance decreased (Investigations) | 1 (1)
Urine calcium oxalate (Investigations) | 2 (8)
Urine protein, quantitative increased (Investigations) | 13 (179)
Venous blood pH decreased (Investigations) | 10 (62)
Venous blood pH increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT03267277/Prot_SAP_000.pdf